CLINICAL TRIAL: NCT06340191
Title: The Influence of Pilates Cueing in Participants With Low Back Pain.
Brief Title: Cueing and Pilates in Low Back Pain
Acronym: PIlatesuja
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJAPIlates1
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain; Pilates Exercise; Pilates, Core Stability; Mind-body Exercise
Keywords: pilates; low back pain; mind-body
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pilates in addition to cueing
  Interventions: Other: Pilates with cueing
- Control group (Active Comparator): Pilates without cueing
  Interventions: Other: Pilates without cueing

INTERVENTIONS:
Other: Pilates with cueing — The Pilates with a cueing component of the intervention involved a specialized approach to Pilates training. Participants in this group underwent an initial phase of training before the main sessions began, which consisted of two smaller group sessions focused on learning explicit verbal and tactile cues. These cues were designed to assist participants in maintaining proper body alignment, engaging specific muscle groups more effectively, and refining their movement techniques to enhance the overall efficacy of the Pilates exercises.
  During the actual Pilates sessions, the instructors, who were certified and brought extensive experience to the program, provided real-time feedback to the participants. This feedback was based on the cueing instructions, aiming to optimize the execution of the Pilates exercises.
  Arms: Intervention group
Other: Pilates without cueing — The Pilates without cueing portion of the study involved participants following the same comprehensive Pilates program as the Pilates with cueing group, with a significant distinction: they did not receive any additional training on cueing. This group engaged in 60-minute Pilates sessions twice a week for 8 weeks, under the supervision of certified and highly experienced Pilates instructors. The program included a variety of exercises, both mat-based and utilizing props, designed to improve participants' physical condition and wellness.
  However, unlike their counterparts in the first group, these participants were not given explicit instructions on how to enhance their body alignment, muscle engagement, or movement techniques through verbal and tactile cues. They performed the Pilates exercises following the standard regimen, without the nuanced guidance and real-time feedback focused on optimizing exercise execution through cueing.
  Arms: Control group

SUMMARY:
The intervention involved two groups participating in supervised Pilates sessions, twice a week for 8 weeks, featuring a mix of mat and props-based exercises. Group 1 received additional cueing training to enhance alignment, muscle engagement, and movement technique, while Group 2 underwent the same Pilates regimen without this cueing component.

DETAILED DESCRIPTION:
The study involved two distinct groups, both of which engaged in Pilates sessions lasting for 60 minutes, held twice a week over eight weeks. These sessions were meticulously overseen by certified Pilates instructors, who brought to the table a wealth of experience. The regimen for the Pilates program was comprehensive, incorporating a blend of exercises performed on mats and with the aid of various props.

The first group, Pilates with cueing, consisted of participants who, before starting the main Pilates sessions, were given additional training. This preliminary phase involved two smaller group sessions where the focus was on learning explicit verbal and tactile cueing. These cues were specifically designed to aid participants in maintaining proper body alignment, engaging the correct muscle groups effectively, and refining their overall movement technique. Throughout the Pilates sessions, instructors provided real-time feedback, aiming to optimize the execution of exercises based on these cues.

The second group, known as Pilates without cueing, participated in an identical Pilates program to that of the first group in terms of the exercises performed, the duration of sessions, and the overall timeframe. However, this group did not receive the preliminary cueing instruction. They performed the Pilates exercises following the same program as the first group but without the added focus on cueing for alignment, muscle engagement, and technique refinement.

ELIGIBILITY:
Inclusion:

* Individuals aged 18 to 65 years.
* Experiencing chronic non-specific low back pain for a minimum of 3 months.
* Ability to participate in supervised exercise programs.
* Absence of medical contraindications for Pilates practice.

Exclusion:

* Vestibular disorders.
* Severe osteoporosis.
* Usual Pilates practitioner.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Low back pain | From baseline to 8 weeks
  Roland Morris Disability Questionnaire (RMDQ): The RMDQ is a self-reported measure widely used to assess physical disability due to lower back pain. It consists of 24 items that reflect the range of activities that might be affected by back pain. The scoring is simple, with higher scores indicating greater disability. This questionnaire is known for its reliability and validity in measuring disability levels in individuals with back pain
Pain report | From baseline to 8 weeks
  Pain was measured using a visual analogue scale (VAS). The VAS consists of a 10-cm line, with the left extremity representing (the absence of pain) and the right extremity indicating (the worse pain devisable). Participants were asked to indicate on the scale their current level of pain being higher values related to more intense pain.

SECONDARY OUTCOMES:
Fear of movement | From baseline to 8 weeks
  The Tampa Scale of Kinesiophobia (TSK) serves as a pivotal tool in assessing the fear of movement or re-injury, particularly among individuals with musculoskeletal pain. It quantifies kinesiophobia (the excessive, irrational fear of physical activity due to apprehensions about pain or further injury) through a questionnaire where respondents rate their agreement with various statements related to movement and pain. This scale is instrumental in identifying psychological barriers to physical activity, enabling healthcare professionals to develop more comprehensive and effective rehabilitation strategies that address both the physical and psychological facets of recovery.
Perceived Stress Scale | From baseline to 8 weeks
  The Perceived Stress Scale (PSS) assesses stress perception over the past month, using a Likert scale in its questions. Scores range from 0 to 40, with higher scores indicating greater perceived stress. It's widely utilized in health research to gauge and manage stress levels.
Pain self-efficacy | From baseline to 8 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) measures an individual's confidence in performing daily activities despite chronic pain, using a scale from 0 to 60, where higher scores signify greater self-efficacy.
Patient Impression of Change | From baseline to 8 weeks
  The Patient Global Impression of Change (PGIC) is a one-item questionnaire that captures a patient's overall perception of change in their condition following treatment, using a 7-point Likert scale from "Very much improved" (1) to "Very much worse" (7). This tool is essential in clinical research for providing a direct, patient-reported outcome measure that reflects the subjective efficacy and impact of interventions. Its simplicity and adaptability across various medical conditions make it a valuable instrument for evaluating patient-centered treatment outcomes.
Body Awareness | From baseline to 8 weeks
  The Body Awareness Questionnaire (BAQ) is a self-report measure designed to assess an individual's attentiveness to internal bodily sensations, encompassing aspects such as recognizing hunger and satiety signals, breathing patterns, and muscle tension. It typically employs a Likert scale for responses, allowing participants to rate their level of agreement with various statements. The BAQ's scoring system is used to quantify the degree of body awareness, with higher scores indicating greater awareness. This tool is valuable in research and clinical settings, particularly in studies of mind-body interventions, psychological well-being, and somatic disorders.

CONTACTS AND LOCATIONS:
Overall Officials: DAVID CRUZ DIAZ, PhD, Principal Investigator — University of Jaén
Locations (1):
- University of Jaen, Jaén, Spain